CLINICAL TRIAL: NCT02169193
Title: Diagnosis of Microaspiration in Intubated Critically Ill Patients: Pepsin vs 99m Technetium
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011_09; 2011-A0140932 (Other: ID-RDB number, ANSM)
Record Dates: First submitted 2014-06-18; First posted 2014-06-23 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Critical Illness
Keywords: microaspiration; mechanical ventilation; enteral feeding; 99m technetium; pepsin
MeSH Terms: conditions — Critical Illness | interventions — nanocis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 99mTc-Rhenium Sulfide Nanocolloid (Experimental): 99mTc-Rhenium Sulfide Nanocolloid
  Interventions: Radiation: 99mTc-Rhenium Sulfide Nanocolloid

INTERVENTIONS:
Radiation: 99mTc-Rhenium Sulfide Nanocolloid — 12 MBq of NanoCis added to 500 ml of enteral feeding
  Other Names: NanoCis

SUMMARY:
Microaspiration of contaminated oropharyngeal secretions and gastric contents frequently occurs in intubated critically ill patients, and plays a major role in the pathogenesis of ventilator-associated pneumonia. Quantitative pepsin measurement in tracheal aspirates would be useful in diagnosing microaspiration of gastric contents in intubated critically ill patients. Technetium 99m labelled enteral feeding is the gold standard for the diagnosis of microaspiration. The investigators hypothesized that tracheal pepsin measurement is a good diagnosis marker of microaspiration compared to the gold standard.

DETAILED DESCRIPTION:
Microaspiration of contaminated oropharyngeal secretions and gastric contents frequently occurs in intubated critically ill patients, and plays a major role in the pathogenesis of ventilator-associated pneumonia Quantitative pepsin measurement in tracheal aspirates would be useful in diagnosing microaspiration of gastric contents in intubated critically ill patients Technetium 99m labelled enteral feeding is the gold standard for the diagnosis of microaspiration. We hypothesized that tracheal pepsin measurement is a good diagnosis marker of microaspiration compared to the gold standard

ELIGIBILITY:
Inclusion Criteria:

* age > or = 18 years
* hospitalised in ICU
* tracheal intubation using a polyvinyl chloride tube and mechanical ventilation
* predictable mechanical ventilation > or = 6 hours after inclusion
* enteral nutrition by a nasogastric tube

Exclusion Criteria:

* refuse to participate to the study
* no informed consent
* pregnant
* contra-indication for enteral nutrition
* tracheotomy
* intubation or re-intubation done in 6 hours preceding the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
incidence of pepsin levels ≥200 ng / ml | from the start to 6 hours after beginning of 99m technetium labelled enteral feeding
  Sensibility and sensitivity of Pepsin for the diagnosis of microaspiration will be determined with regard to 99m technetium (gold standard).

SECONDARY OUTCOMES:
likelihood ratio of pepsin of microregurgitation | from the start to 6 hours after beginning of 99m technetium labelled enteral feeding
  Sensibility and sensitivity of Pepsin for the diagnosis of microregurgitation will be determined with regard to 99m technetium.
likelihood ratio of pepsin of microaspiration | from the start to 6 hours after beginning of 99m technetium labelled enteral feeding
  positive and negative predictive values, positive and negative likelihood ratio of pepsin for the diagnosis of microaspiration compared to the 99m technetium (gold standard)
Youden Index | from the start to 6 hours after beginning of 99m technetium labelled enteral feeding
  Youden Index and ROC curve analysis of the Pepsin as a marker for the diagnosis of microaspiration compared to the 99m Technetium (gold standard)
ROC curve | from the start to 6 hours after beginning of 99m technetium labelled enteral feeding
  Youden Index and ROC curve analysis of the Pepsin as a marker for the diagnosis of microaspiration compared to the 99m Technetium (gold standard)

CONTACTS AND LOCATIONS:
Overall Officials: Saad Nseir, MD, PhD, Principal Investigator — Univ Hosp of Lille, France
Locations (1):
- ICU, Calmette Hospital, University Hospital of Lille, Lille, France